CLINICAL TRIAL: NCT04100993
Title: Growing up on Non-invasive Ventilation: Assessment of Multisystem and Autonomic Complications of Neuromuscular and Neurological Disorders in Young Adults
Brief Title: Multisystem and Autonomic Complications of NMD on Long-term NIV
Status: Completed | Type: Observational
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 266270
Record Dates: First submitted 2019-07-31; First posted 2019-09-24 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Neuromuscular Diseases; Neurologic Disorder
MeSH Terms: conditions — Neuromuscular Diseases; Nervous System Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient group: 60 participants ≥16 years of age with a confirmed diagnosis of a childhood-onset NMD
  Interventions: Other: No intervention used
- Exploratory reference group: 20 healthy adults ≥16 years of age
  Interventions: Other: No intervention used

INTERVENTIONS:
Other: No intervention used — No intervention used

SUMMARY:
This exploratory observational study evaluates autonomic function using measures including heart rate variability in adults with childhood-onset neuromuscular and neurological disorders (NMD) who use non-invasive ventilation (NIV) as part of their long-term care. Autonomic function will be correlated with measures of symptom burden, disease severity and complications.

DETAILED DESCRIPTION:
Childhood-onset neuromuscular and neurological disorders (NMD) are a diverse group of rare conditions in which muscle function is significantly impaired. Due to progress in NMD management over recent decades, particularly the use of non-invasive ventilation (NIV) to treat chronic respiratory failure, many individuals are surviving into adulthood and even middle age. However, older individuals are developing potentially fatal complications related to the heart e.g. sudden cardiac death, gastrointestinal (GI) tract and increasing dependence on NIV.

Previous studies largely in children and adolescents suggest individuals with NMD may develop problems of the autonomic nervous system (ANS), a network of nerves vital to controlling the body's short-term responses to internal and external stimuli. It is likely some complications of NMD are related to ANS abnormalities.

This will be an exploratory observational study using a cross-sectional design in which non-invasive tools will be used to evaluate autonomic function during wake and sleep. Individuals over 16 years of age with a confirmed NMD diagnosis will be recruited. Derived parameters of autonomic function including heart rate variability will be compared to values from an exploratory reference group of age- and sex-matched healthy adults. Autonomic function will also be correlated to measures of symptom burden, complications, quality of life and disease severity. Qualitative methods will be used to further evaluate the experience and perceptions of adults with NMD in making decisions about their personal and medical care, which become more complex with increasing age and disease severity.

ELIGIBILITY:
Inclusion Criteria:

Patient group:

* Age ≥16 years
* Confirmed diagnosis of childhood-onset NMD
* Able and willing to provide informed consent
* Requires non-invasive ventilation on an intermittent or continuous basis to manage respiratory failure

Reference group:

* Age ≥16 years
* No significant co-morbidities
* Not on any regular medications
* Able and willing to provide informed consent

Exclusion Criteria:

* Inability to travel to hospital site
* Clinical instability or acute deterioration requiring hospitalisation or changes to medication in the previous 4 weeks
* A female of child-bearing potential who is pregnant or intends to become pregnant during study involvement

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a relevant NMD who attend adult Sleep and Ventilation services at the study site will be identified by the direct care team.
  Healthy age- and sex-matched adults from the local community will be invited to participate by the research team.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2021-05-20 (Actual)

PRIMARY OUTCOMES:
Heart rate variability (HRV) | 1 day
  HRV will be analysed in time and frequency domains from short-term (5 minute) artefact free ECG recordings. Normal parameters will be determined from an age- and sex-matched exploratory reference group of healthy adults.

SECONDARY OUTCOMES:
Baroreflex sensitivity (BRS) | 1 day
  BRS will be analysed in time and frequency domains from short-term (5 minute) artefact free blood pressure recordings. Normal parameters will be determined from an age- and sex-matched exploratory reference group of healthy adults. This will be measured only in the patient participant group.
Composite Autonomic Symptom Scale 31 questionnaire | 1 day
  Composite Autonomic Symptom Scale 31 questionnaire (COMPASS 31) is a validated questionnaire for quantitative assessment of autonomic symptoms, based on the original Autonomic Symptom Profile. The 31 questions are divided into seven domains (orthostatic intolerance, vasomotor, secretomotor, gastrointestinal, bladder and pupillomotor). The raw score from each domain is multiplied by a weight index to give a total score with a maximum score of 100 (minimum score 0). Higher scores indicate greater symptom burden.
Sydney Swallow Questionnaire | 1 day
  The Sydney Swallow Questionnaire (SSQ) is a validated self-reported inventory of 17 questions measuring symptomatic severity of oral-pharyngeal dysphagia using 16 visual analogue scales (VAS) and one question scored on a Likert scale (0-5) to rate swallowing difficulty and symptoms of dysphagia and aspiration in a range of situations. Each VAS measures 100mm; the raw scores from these are added to the weighted score of the additional question to make the total possible raw score 1700 when the scores are added. Higher scores indicate greater symptom burden. This will be measured only in the patient participant group.
The European Quality of Life - 5 Dimensions questionnaire | 1 day
  The European Quality of Life - 5 Dimensions questionnaire (EQ-5D-5L) is a standardised instrument developed by the EuroQol Group as a measure of health-related quality of life that can be used in a wide range of health conditions and treatments. The EQ-5D-5L consists of a descriptive system comprising five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression, each with 5 levels of severity. An EQ visual analogue scale then asks patients how they feel on the day of the visit. A unique health state is defined by sequentially combining the indicated level in each of the 5 dimensions. This will be measured only in the patient participant group.
Patient Assessment of Constipation Symptoms questionnaire | 1 day
  The Patient Assessment of Constipation Symptoms questionnaire (PAC-SYM) is a symptom inventory which measures specific symptoms of constipation in adults. It consists of a 12-item measure of patient's experience of symptoms and symptom severity. The score of each question is given equal weight and domain and total scores can be calculated by summing the relevant scores and dividing by the number of non-missing items. This will be measured only in the patient participant group.
Individualized Neuromuscular Quality of Life Questionnaire | 1 day
  The Individualized Neuromuscular Quality of Life Questionnaire (INQoL) is a validated muscle disease specific measure use to assess health-related quality of life of adult patients with acquired or congenital neuromuscular diseases, developed from the experiences of patients with muscle disease. It consists of 45 questions within 10 sections. Four sections focus on the impact of key muscle disease symptoms; five assess at the degree and importance of impact muscle disease has on particular areas of life; one section asks about positive and negative effects of treatment. The questionnaire allows for variations in individual characteristics that influence quality of life. The scoring of the INQoL generates a profile and combining weighted scores of each domain produces a total score from 0 to 100, with higher scores indicate greater impact of disease. This will be measured only in the patient participant group.
Severe Respiratory Insufficiency quality of life tool | 1 day
  The severe Respiratory Insufficiency quality of life tool (SRI)is a validated questionnaire assessing health-related quality of life in patients with respiratory failure on home ventilation. It consists of seven subscales covering 49 items rated on a 5-point Likert scale: respiratory complaints, physical functioning, attendant symptoms and sleep, social relationships, anxiety, psychological wellbeing and social functioning. After transformation and weighting of raw scores, a total score between 0 and 100 is calculated. Higher values indicate a better health-related quality of life. This will be measured only in the patient participant group.
Forced Expiratory Volume in 1 second (FEV1) | 1 day
  The best of 3 attempts obtained through standard Spirometric assessment will be used to obtain FEV1 (L) in the patient participant group.
Forced Expiratory Volume (FVC) | 1 day
  The best of 3 attempts obtained through standard Spirometric assessment will be used to obtain FVC (L) in the patient participant group.
Ratio of FEV1/FVC | 1 day
  The values obtained from standard Spirometric assessment will be used to determine FEV1/FVC ratio in the patient participant group.
Peak cough flow | 1 day
  Using a standard peak flow meter, peak cough flow will be recorded in L/min the patient participant group.
Sniff nasal inspiratory pressure | 1 day
  Sniff nasal inspiratory pressure (SNIP) in each nostril will be recorded in the patient participant group.
Brain natriuretic peptide | 1 day
  Serological brain natriuretic peptide (BNP) will be obtained through venepuncture in the patient participant group.
Troponin-I | 6 months
  Serological troponin will be obtained through venepuncture in the patient participant group.
Arterialised blood gas tensions | 1 day
  Standard blood gas tensions will be obtained from earlobe puncture in the patient participant group.
Colon transit study | 1 day
  Single abdominal x-ray to evaluate number of retained radiopaque markers 5-days after oral ingestion in the patient participant group.
Themes describing patient perceptions of experiences and needs in complex clinical and non-clinical decision making | 1 hour
  Inductive thematic analysis of individual interviews to provide qualitative data in the patient participant group.
Weight | 1 day
  Measured using calibrated scales in kilograms
Height | 1 day
  Measured using calibrated scales in centimetres
Body Mass Index | 1 day
  Calculated using the formula BMI = weight(kg)/[height(m)]2
Nocturnal transcutaneous carbon dioxide | 1 day
  Nocturnal transcutaneous carbon dioxide will be measured overnight in kilopascals (kPa)
Cardiac function | 1 day
  Standard transthoracic echocardiogram will be performed in the patient participant group to assess cardiac function

CONTACTS AND LOCATIONS:
Overall Officials: Anita K Simonds, MD MBBS, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust
Locations (1):
- Royal Brompton Hospital, London, United Kingdom